CLINICAL TRIAL: NCT00611104
Title: Evaluation of the Aromatase Inhibition Potential of Standardized Grape Extract
Brief Title: Studying the Effect of Freeze-Dried Table Grape Powder on Blood Estrogen Levels in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC0536; CDR0000581219 (Other: Sponsor Protocol Number); 06-002061 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2008-02-07; First posted 2008-02-08 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: standardized freeze-dried table grape powder
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Studying samples of blood and urine in the laboratory from participants receiving freeze-dried table grape powder may help doctors understand the effect of this drug on blood estrogen levels.

PURPOSE: This clinical trial is studying the effect of freeze-dried table grape powder on blood estrogen levels in postmenopausal women.

DETAILED DESCRIPTION:
OBJECTIVES:

* To measure the change in levels of plasma estrone (E1), estradiol, E1-conjugates, and E1-sulfates in postmenopausal women after 6 weeks of daily ingestion of 94 grams of freeze-dried table grape powder.
* To conduct bioavailability research on the freeze-dried table grape powder in humans through the analysis of participants' blood and urine samples.

OUTLINE: Participants receive oral freeze-dried table grape powder once daily on days 1-42 in addition to their usual diet. Treatment continues in the absence of toxicity.

Participants undergo blood sample collection at baseline, periodically after the first dose, and on the last day of the study for pharmacokinetic and bioavailability analysis. Samples are examined by mass spectrometry to measure plasma levels of estrone (E1), estradiol, E1-conjugates, E1-sulfates, testosterone, and androstenedione. Participants also undergo spot urine collection and weight and height measurement periodically during study.

Participants complete food diaries on days 1-3, 21-23, and 40-42 to assess their intake of grapes, grape juice, and red wine and to examine the constancy of their caloric intake over the course of the study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Participant in the Mayo Mammography Health Study

  * Has consented to provide baseline mammogram for digitization

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Female
* Postmenopausal (defined as women who have had both ovaries removed or no menstrual period for at least 12 consecutive months)
* Able to give informed consent and complete food records alone or with assistance
* Willing to provide research blood and urine samples
* Must be a non-smoker
* Willing to maintain current weight
* No history of breast ductal carcinoma in situ or any other cancer, except basal cell or squamous cell skin cancer or lobular carcinoma in situ
* No history of allergic or other adverse reaction to grapes
* No history of diabetes or glucose intolerance

PRIOR CONCURRENT THERAPY:

* No concurrent hormone therapy, including estradiol, estrone, or progestins

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PATIENT CHARACTERISTICS:
  * ECOG performance status 0-1
  * Female
  * Postmenopausal (defined as women who have had both ovaries removed or no menstrual period for at least 12 consecutive months)
  * Able to give informed consent and complete food records alone or with assistance
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-08-04 (Actual); Primary Completion 2014-08-22 (Actual); Study Completion 2014-08-22 (Actual)

PRIMARY OUTCOMES:
Serum levels of plasma estrone (E1), estradiol, E1-conjugates, and E1-sulfates
Bioavailability of the freeze-dried table grape powder in humans

CONTACTS AND LOCATIONS:
Overall Officials: Janet E. Olson, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States